CLINICAL TRIAL: NCT04865575
Title: Systems Pharmacology Approach to Uncontrolled Pediatric Asthma (SysPharmPediA)
Brief Title: Systems Pharmacology Approach to Uncontrolled Pediatric Asthma
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University of Maribor, Maribor, Slovenia. (Unknown); University Children's Hospital, University of Regensburg, Regensburg, Germany (Unknown); Universidad de La Laguna, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain. (Unknown); University of the Basque Country (UPV/EHU) (Other); Hospital Universitario Donostia, San Sebastián, Spain. (Unknown); Instituto de Salud Carlos III (Other Government); Utrecht University, Utrecht, the Netherlands. (Unknown); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Prof. dr. A.H. Maitland-van der Zee, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL55788.041.15
Record Dates: First submitted 2021-04-21; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Pediatric Asthma; Uncontrolled Asthma
Keywords: Systems Pharmacology; Omics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, feces, saliva, nasal swabs and exhaled breath.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- controlled asthmatics: moderate-to-severe asthmatic children with good asthma control
- uncontrolled asthmatics: moderate-to-severe asthmatic children with poor asthma control / recurrent exacerbations

SUMMARY:
Background:

Asthma is a heterogeneous respiratory disease and the most common chronic disease in children. A small subset of children has continuous poor asthma control despite appropriate adherence to asthma medication. There is a clinical need to identify these children as early as possible to optimize treatment and/or to find therapeutic alternatives. Therefore, the "Systems Pharmacology approach to uncontrolled Pediatric Asthma" (SysPharmPediA) study was set up.

Objective:

To establish a cohort of pediatric moderate-to-severe uncontrolled and controlled patients with asthma in order to investigate pathophysiological mechanisms underlying uncontrolled moderate-to-severe asthma in children on maintenance treatment, using a multi-omics systems medicine approach.

Methods:

In this multicenter observational case-control study, moderate-to-severe asthmatic children (n=145, age 6-17 years), were included in specialized hospitals in four European countries (Netherlands, Germany, Spain and Slovenia). Recruited subjects were selected based on good asthma control (controlled asthmatics, n=54) or poor asthma control / recurrent exacerbations (uncontrolled asthmatics, n=91). Comprehensive details concerning demographics, current and past patient/family history and clinical characteristics were collected. In addition, systems-wide omics layers, including epi(genomics), transcriptomics, microbiome, proteomics and metabolomics will be evaluated from multiple collected, relatively non-invasive, samples of from the recruited individuals, such as: blood, feces, saliva, nasal swabs and exhaled breath. Follow-up visits were performed 6 and 12 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

General:

* Between 6-17 years of age
* Doctor diagnosis of asthma

In addition to the general criteria, a case with uncontrolled asthma (case group A) should meet:

* Asthma treatment Global INitiative of Asthma (GINA) step 3 or higher

  ≥ 1of the following criteria (based on the guideline 'Childhood Asthma' of the section paediatric pulmonology of the Dutch Society of Paediatricians, 2007):
* Frequent exacerbations requiring OCS use (≥1 in the past year) and/or
* Severe exacerbations requiring hospitalization or ER visits in the past year and/or
* ACQ/ACT scores indicating uncontrolled asthma

In addition to the general criteria, a case with an acute exacerbation (case group B) should meet:

* Asthma treatment Global INitiative of Asthma (GINA) step 2 or higher
* Current severe asthma exacerbation requiring hospitalization

In addition to the general inclusion criteria, a control (controlled asthma) should meet the following criteria:

* Asthma treatment Global INitiative of Asthma (GINA) step 3 or higher
* Lack of severe exacerbations requiring OCS use or hospitalizations or ER visits in the past year
* ACQ/ACT scores indicating well controlled asthma or few reported asthma symptoms during asthma checks in the past year.

Exclusion Criteria:

* Recent use of a course of antibiotics (< 1 month). This will affect the microbiome analyses.

A patient can be re-screened 1 month after the use of the antibiotic treatment has finished.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Four tertiary care centers from four European countries (the Netherlands, Germany, Spain, and Slovenia) recruited 145 asthmatic children and adolescents (6-17 years old). All centers obtained approval from their local medical ethics committee (ethics committee of University Regensburg, Germany (18-1034-101); Clinical Research Ethics Committee of the Basque Country, Spain (PI2015075 (SO)); Medical Ethics Committee of the University Medical Center Utrecht (UMC Utrecht), Utrecht, the Netherlands (NL55788.041.15); National Medical Ethics Committee, Slovenia (0120-569/2017/4)) and written informed consents were collected from the parents/caregivers and/or the recruited children when appropriate.
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Saliva and stool microbiome | Baseline
  Differences in 16S rRNA microbial α- and ß- diversities between cases and controls
Exhaled breath metabolome | Baseline
  Differences in presence and levels of volatile organic compounds between cases and controls

OTHER OUTCOMES:
Age | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  Age in years
Sex | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  Female/Male
BMI | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  kg/m2
Uncontrolled asthma | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  according to the Asthma Control Test (ACT) questionnaire (<19 score) and frequent exacerbation within the past 12 months (>n of exacerbation in the past 12 months
Exacerbations | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  Exacerbation requiring OCS use, hospitalization or ER visit
Spirometry | Baseline
  FEV1 (L, percent predicted value)
Pediatric Asthma Quality of Life Questionnaire (PAQLQ) | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  Questionnaire including 23 questions in 3 domains (symptoms, activity limitation, emotional function) and a 7-point scale (7 = not bothered at all; 1 = extremely bothered)
Atopy | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  Questionnaire on history of allergic diseases
Current asthma medication intake | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  ICS: inhaled corticosteroids, LTRA: leukotriene antagonist, SABA: short-acting beta agonist, LABA: long-acting beta agonist, OCS: oral corticosteroids, Omalizumab, Mepolizumab
Asthma severity | Baseline (+ follow-up at 6 and 12 months after baseline inclusion)
  Asthma Control Test (ACT)

CONTACTS AND LOCATIONS:
Locations (6):
- University Regensburg, Regensburg, Germany
- Utrecht University, Utrecht, Netherlands
- University of Maribor, Maribor, Slovenia
- Spain (2):
  - University of the Basque Country, San Sebastián
  - Universidad de La Laguna, Santa Cruz de Tenerife
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
In case other researchers are interested to work with data that is collected within SysPharmPediA; we kindly request to contact the PI of the study (Prof. dr. A.H. Maitland-van der Zee - a.h.maitland@amsterdamumc.nl)
  1. The PIs will refer to an up-to-list of planned publications, which includes ongoing and planned analysis work from SysPharmPediA partners and from those granted access to specific data, to determine potential duplication of work.
  2. To understand and draw sound scientific results those groups planning to work on SysPharmPediA data should engage with the SysPharmPediA members who have generated the data in question.
  3. A summary of the Data Analysis Plan (DAP) must be attached to the data access request form.
  4. If the analysis deviates substantially from the summary DAP or provides results which the SysPharmPediA group feel mis-represent the data, the SysPharmPediA group may raise an objection with the publication concerned.